CLINICAL TRIAL: NCT04318899
Title: Predictors of Clinical Course and Treatment Response in Patients Having Received Dialectical Behaviour Therapy Delivered by Clinical Units in the Norwegian Network for Clinical Evaluation and Quality in DBT Programmes
Brief Title: Predictors of Clinical Course and Treatment Response in DBT Programmes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other); St. Olavs Hospital (Other); Sykehuset Ostfold (Other); University of Oslo (Other); Nordlandssykehuset HF (Other)
Responsible Party: Principal Investigator, Lars Mehlum, Professor dr med, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1247/REK sør-øst
Record Dates: First submitted 2020-03-04; First posted 2020-03-24 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Self Harm; Borderline Personality Disorder
Keywords: self harm; dialectical behaviour therapy; borderline personality disorder; emotional dysregulation
MeSH Terms: conditions — Self-Injurious Behavior; Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dialectical Behaviour Therapy (Experimental): Dialectical Behavior Therapy, delivered for 20 weeks for adolescents (DBT-A) or 52 weeks for adults (standard DBT.
  Interventions: Behavioral: Dialectical Behaviour Therapy adapted for adolescents (DBT-A); Behavioral: Dialectical Behaviour Therapy - Standard version (DBT)

INTERVENTIONS:
Behavioral: Dialectical Behaviour Therapy adapted for adolescents (DBT-A) — DBT developed by Marsha Linehan (Linehan 1993a; 1993b) and adapted for adolescents (DBT-A) by Miller, Rathus & Linehan, 2007 consisting of 20 weeks of weekly individual therapy (60 minutes), multifamily skills training (120 minutes), family therapy sessions as needed and telephone coaching outside therapy sessions.
Behavioral: Dialectical Behaviour Therapy - Standard version (DBT) — DBT developed by Marsha Linehan (Linehan 1993a, 1993 b) consisting of 1 weekly session of individual therapy (60 minutes), 1 weekly session of skills training (120 minutes), and telephone coaching with individual therapists outside therapy sessions as needed.

SUMMARY:
The project is a collaboration between The National Centre for Suicide Research and Prevention (NSSF) and clinical units with Dialectical Behaviour Therapy (DBT) programmes. A methodological and technological platform has been established that enables clinicians to deliver high quality treatments over extended periods of time, to evaluate their own performance and productivity and to report it in a uniform and systematic way that will enable comparison across clinical settings and programmes. The collected data constitute the basis for conducting the clinical study with the overall aim to study predictors of the clinical course and treatment response in patients admitted to DBT programmes in Norway.

DETAILED DESCRIPTION:
The aim of the project is to collect data from systematic and uniform clinical assessments to study predictors of the clinical course and treatment response in patients admitted to and treated in clinical units delivering Dialectical Behaviour Therapy in Norway.

Aims and research questions:

The study will address the following main research questions:

1. Which patient characteristics (sociodemographic variables, psychiatric diagnoses/comorbidities, previous suicidal and self-harming behaviour, previous treatment history), predict a favourable clinical course and treatment response?
2. Which factors mediate the clinical change in key outcomes such as a) target symptom levels (depression, hopelessness, suicidal ideation, borderline symptoms etc.), b) function levels (emotion regulation capacity, use of coping skills, social functioning, occupational / academic performance level etc.), c) problem behaviours (suicide attempts, non-suicidal self-harm, substance abuse, eating disorder symptoms etc.), d) global functioning and e) the use of emergency treatment services.
3. What are significant moderators of treatment response with respect to key clinical outcomes (mentioned above)?
4. Which of the treatment modalities are evaluated as the most salient and helpful by patients who receive the treatment according to their age, gender, psychiatric diagnoses and previous treatment history?

Methods:

A uniform protocol for psychiatric diagnostics and clinical assessment of patients who receive treatment at the participating clinical units will be used. Since some participating clinical units will treat adult patients and some will treat children and adolescents, the protocol will offer assessment instrument suitable for the specific age group whenever this is relevant. The evaluation system includes assessments at baseline before treatment starts, evaluation at several time points during the treatment period, at termination of treatment and at follow-up. Assessments will be made both through interviews and ratings made by therapists and through self-report from patients.

Self-reports will be filled out electronically by patients, on tablets stationed at each participating clinical unit. At intervals patients will also provide self-rated information on dimensions such as emotions, cognitions and impulsive behaviour several times per day through a mobile app developed specifically for the purpose, so-called Ecological Momentary Assessment (EMA). Interview data and ratings will be entered into the database by each clinician to tablets in a similar fashion as self-report data from patients.

ELIGIBILITY:
Inclusion Criteria:

* History of repeated deliberate self harm
* Satisfies criteria of Diagnostic and Statistical Manual (DSM-IV) Borderline Personality Disorder as measured by Structured Clinical Interview for the DSM (SCID-II) in addition to the self-destructive criterion.

Exclusion Criteria:

* Psychotic disorders
* Anorexia Nervosa
* Substance dependence disorder
* Mental retardation (IQ less than 70)
* Asperger syndrome/autism

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-harm behaviour | 4 weeks
  Number of self-harm episodes (split on suicide attempts and non-suicidal self-harm)
Suicidal Ideation (adolescents) | 2 weeks
  Suicidal Ideation Questionnaire (SIQ-Jr). Min=0, Max=90. Higher scores indicate worse outcome
Depressive symptoms | 1 week
  MADRS (Montgomery Asberg Depression Rating Scale).Min=0, Max=60. Higher scores indicate worse outcome
Suicidal Ideation (adults) | 4 weeks
  Beck Scale for Suicidal Ideation (BSS). MIn=0, Max=38. Higher scores indicate worse outcome
Depressive symptoms (adolescents) | 1 week
  Moods and Feelings Questionnaire (MFQ). Min=0, Max=26. Higher scores indicate worse outcome
Depressive symptoms (adults) | 1 week
  Beck Depression Inventory (BDI). Min=0, Max=63. Higher scores indicate worse outcome

SECONDARY OUTCOMES:
Borderline Symptoms | 1 week
  Borderline Symptom List (BSL-23). Min=0, Max=92. Higher scores indicate more symptoms.
Hopelessness | 1 week
  Beck Hopelessness Scale (BHS). Min=0, Max=20. Higher scores indicate more hopelessness.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Mehlum, MD PhD, Principal Investigator — University of Oslo
Locations (5):
- Norway (5):
  - Søndre Oslo DPS/Oslo Universitetssykehus HF, Oslo, Oslo County
  - Moss DPS/Østfold sykehus HF, Moss
  - Psykiatrisk senter ytre Helgeland/Helgelandssykehuset HF, Sandnessjøen
  - Bjerketun behandlingshjem/Vestreviken HF, Sandvika
  - BUP Lian/St Olavs Hospital HF, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linehan, M.M. (1993a). Cognitive-behavioral treatment of borderline personality disorder. New York: Guilford Press
- [Background] Linehan, M.M. (1993b). Skills training manual for treating borderline personality disorder. New York: Guilford Press
- [Background] Miller, A.L., Rathus J.H., Linehan, M.M. (2007). Dialectical behavioral therapy with suicidal adolescents. New York: Guilford Press